CLINICAL TRIAL: NCT07272213
Title: Evaluation of the Effects of Thyroid-Stimulating Hormone (TSH) Levels in Pregnancy on Depression, Anxiety, and Sexual Function
Brief Title: Thyroid-Stimulating Hormone Levels in Pregnancy and Their Association With Depression, Anxiety, and Sexual Function
Acronym: TSH-MIND
Status: Recruiting | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Havva Betül Bacak, Specialist in Obstetrics and Gynecology, Gaziosmanpasa Research and Education Hospital
Other Study IDs: GOPKAD-TSH-DEP-2025
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Thyroid Disorders Complicating Pregnancy; Maternal Depression in Pregnancy, Unspecified Trimester; Anxiety Disorder, Unspecified; Sexual Dysfunction, Unspecified
Keywords: Thyroid disorders complicating pregnancy; Maternal depression in pregnancy, unspecified trimester; Anxiety disorder, unspecified; Sexual dysfunction, unspecified
MeSH Terms: conditions — Anxiety Disorders; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TSH ≤2.5 Group: Participants in this cohort have serum TSH levels ≤2.5 mIU/L. No intervention will be administered. Participants will undergo psychometric evaluation using the Beck Depression Inventory (BDI), Beck Anxiety Inventory (BAI), the Arizona Sexual Experience Scale (ASEX), and the YKK-13 Quality of Life Scale. The purpose is to assess psychological and sexual function outcomes in relation to normal-range TSH levels.
- TSH >2.5 Group: Participants in this cohort have serum TSH levels >2.5 mIU/L. No intervention will be administered. Participants will complete the same psychometric assessments (BDI, BAI, ASEX, YKK-13). This group will allow comparison of psychological, anxiety-related, sexual function, and quality-of-life outcomes associated with elevated TSH levels during pregnancy.

SUMMARY:
This prospective, single-center, observational cross-sectional study aims to evaluate the relationship between thyroid-stimulating hormone (TSH) levels and psychological as well as sexual health outcomes during pregnancy. Pregnant individuals will undergo psychometric assessment using the Beck Depression Inventory (BDI), Beck Anxiety Inventory (BAI), the Arizona Sexual Experience Scale (ASEX), and the YKK-13 Quality of Life Scale. The study will investigate whether maternal TSH levels are associated with depression, anxiety, sexual function, and overall quality of life scores.

Eligible participants will be pregnant women aged 18-45 years with a singleton pregnancy of at least 6 weeks, who are literate and have provided informed consent. Individuals with a prior psychiatric history, multiple gestation, or existing systemic or endocrine diseases will be excluded. The primary endpoint of the study is to determine the association between TSH levels and psychometric scale scores during pregnancy.

DETAILED DESCRIPTION:
Pregnancy is a period characterized by significant physiological, hormonal, and psychological changes that may influence maternal well-being. Thyroid-stimulating hormone (TSH) plays a central role in endocrine regulation during pregnancy, and alterations in thyroid function have been associated with mood disorders, anxiety symptoms, and changes in sexual function. Despite emerging evidence suggesting a link between thyroid status and maternal mental health, the relationship between TSH levels and psychological outcomes during pregnancy remains insufficiently explored.

This prospective, single-center, observational cross-sectional study aims to systematically evaluate the association between maternal TSH levels and psychometric parameters, including depression, anxiety, sexual function, and quality of life. Participants will be assessed using validated instruments: the Beck Depression Inventory (BDI), Beck Anxiety Inventory (BAI), the Arizona Sexual Experience Scale (ASEX), and the YKK-13 Quality of Life Scale. Blood samples will be collected to measure serum TSH levels, and questionnaire scores will be obtained during routine prenatal follow-up visits.

The study population will consist of pregnant women aged 18-45 years with a singleton pregnancy of at least six weeks' gestation. Individuals with a history of psychiatric disorders, multiple gestations, or systemic/endocrine diseases will be excluded to minimize confounding factors. Data will be analyzed to determine whether variations in TSH levels are correlated with psychometric outcomes, and to better understand the potential role of thyroid function in maternal psychological and sexual health.

The ultimate goal of this research is to provide clinical insight into how thyroid function may influence mental and sexual well-being during pregnancy, thereby supporting early identification and management of at-risk pregnant individuals.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women aged 18-45 years

Singleton pregnancy

Gestational age ≥ 6 weeks

Literacy and ability to provide informed consent

Availability of a TSH result obtained within the past 4 weeks

Cognitive ability sufficient to complete the psychometric questionnaires (Beck Depression Inventory, Beck Anxiety Inventory, ASEX, and YKK-13 Quality of Life Scale)

Exclusion Criteria:

Multiple pregnancy

Previously diagnosed psychiatric disorder or active use of antidepressant/ anxiolytic medication

Current treatment for thyroid disease

History of thyroid surgery

Major systemic illness or significant obstetric complications

Age under 18 years or inability to provide informed consent

Inability to complete the questionnaires adequately (missing or invalid data)

Rationale:

Multiple pregnancies are excluded because they differ significantly from singleton pregnancies in terms of hormonal profile, obstetric risks, and psychological stress levels. This exclusion aims to ensure a homogeneous study population.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of pregnant women aged 18-45 years who are receiving routine prenatal care at SBÜ Gaziosmanpaşa Training and Research Hospital. Eligible participants will have a singleton pregnancy of at least 6 weeks' gestation, a recent TSH measurement obtained within the past 4 weeks, and sufficient cognitive ability to complete standardized psychometric assessments. Individuals with multiple gestation, diagnosed psychiatric disorders, thyroid disease requiring treatment, major systemic illness, or obstetric complications will be excluded to ensure a homogeneous cohort.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Association Between TSH Levels and Psychometric Scale Scores | At enrollment (single visit).
  To evaluate the relationship between maternal TSH levels (≤2.5 mIU/L vs. >2.5 mIU/L) and psychological outcomes measured by the Beck Depression Inventory (BDI), Beck Anxiety Inventory (BAI), the Arizona Sexual Experience Scale (ASEX), and the YKK-13 Quality of Life Scale. The primary endpoint is the difference in psychometric scores between the two TSH groups and the correlation between serum TSH levels and these scores.

CONTACTS AND LOCATIONS:
Overall Officials: havva betül bacak, md, Principal Investigator — SBÜ Gaziosmanpaşa Training and Research Hospital
Locations (1):
- SBÜ Gaziosmanpaşa Training and Research Hospital, Istanbul, Gaziosmanpaşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No